CLINICAL TRIAL: NCT07000773
Title: Trapezius Activation During Bilateral Scapular Retraction With Shoulder External Rotation: The Incorporation of Knetic Chain and Unstable Surface
Brief Title: Trapezius Muscle Activation During Bilateral Scapular Retraction and Shoulder External Rotation Under Kinetic Chain and Unstable Surface Conditions
Acronym: BSR-SER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Gamze Çobanoğlu Demirkan, Research Assistant, PhD, Physiotherapist, Department of Physiotherapy and Rehabilitation, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Gazi-BSR-SER
Record Dates: First submitted 2025-05-22; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
Keywords: scapular muscle activation; Electromyography; Kinetic Chain; Scapular Retraction; Trapezius; Unstable Surface
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a randomized crossover study where each participant performs the Bilateral Scapular Retraction with Shoulder External Rotation (BSR-SER) exercise under multiple conditions. The exercise is performed on both stable and unstable surfaces and in different lower extremity positions (standing, lunge, and squat). Each participant acts as their own control by completing all exercise conditions in a randomized order. Electromyographic (EMG) activity of the trapezius muscles is measured during each condition to assess muscle activation patterns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Standing on Stable Surface (Experimental): Participants perform the bilateral scapular retraction with shoulder external rotation (BSR-SER) exercise in a standing position on a stable surface using resistance bands.
  Interventions: Behavioral: Bilateral Scapular Retraction with Shoulder External Rotation (BSR-SER) Exercise
- Standing on Unstable Surface (Experimental): Participants perform the BSR-SER exercise in a standing position on an unstable surface (BOSU®) using resistance bands.
  Interventions: Behavioral: Bilateral Scapular Retraction with Shoulder External Rotation (BSR-SER) Exercise
- Lunge Position on Stable Surface (Experimental): Participants perform the BSR-SER exercise in a lunge position on a stable surface using resistance bands. Knee and trunk angles are standardized.
  Interventions: Behavioral: Bilateral Scapular Retraction with Shoulder External Rotation (BSR-SER) Exercise
- Lunge Position on Unstable Surface (Experimental): Participants perform the BSR-SER exercise in a lunge position on an unstable surface (BOSU®) using resistance bands. Knee and trunk angles are standardized.
  Interventions: Behavioral: Bilateral Scapular Retraction with Shoulder External Rotation (BSR-SER) Exercise
- Squat Position on Stable Surface (Experimental): Participants perform the BSR-SER exercise in a squat position on a stable surface using resistance bands. Knee and trunk angles are standardized.
  Interventions: Behavioral: Bilateral Scapular Retraction with Shoulder External Rotation (BSR-SER) Exercise
- Squat Position on Unstable Surface (Experimental): Participants perform the BSR-SER exercise in a squat position on an unstable surface (BOSU®) using resistance bands. Knee and trunk angles are standardized.
  Interventions: Behavioral: Bilateral Scapular Retraction with Shoulder External Rotation (BSR-SER) Exercise

INTERVENTIONS:
Behavioral: Bilateral Scapular Retraction with Shoulder External Rotation (BSR-SER) Exercise — Participants perform the Bilateral Scapular Retraction with Shoulder External Rotation (BSR-SER) exercise using a resistance band. The exercise is conducted under various conditions including stable and unstable surfaces (using BOSU® balance trainer) and in three different lower limb positions: standing, lunge, and squat. Each condition is randomized, and participants complete all conditions in a crossover design. The intervention aims to evaluate trapezius muscle activation patterns during these exercises using surface electromyography (EMG).

SUMMARY:
This study aims to investigate the effects of performing the Bilateral Scapular Retraction with Shoulder External Rotation (BSR-SER) exercise under kinetic chain involvement and unstable surface conditions on trapezius muscle activation. Surface electromyography (EMG) will be used to assess the activity levels of the upper, middle, and lower trapezius muscles. The goal is to determine whether integrating kinetic chain elements and instability can optimize muscle activation patterns in healthy individuals during a commonly used scapular rehabilitation exercise.

DETAILED DESCRIPTION:
Maintaining muscular balance among the scapular stabilizers is crucial for optimal shoulder function. The Bilateral Scapular Retraction with Shoulder External Rotation (BSR-SER) exercise is frequently used in clinical rehabilitation to activate the lower trapezius while minimizing upper trapezius activity. Although this exercise is widely practiced, the effects of performing it under kinetic chain conditions (such as squat and lunge positions) and on an unstable surface have not been thoroughly explored.

This study will examine how adding kinetic chain involvement and instability influences the electromyographic activity of the upper trapezius (UT), middle trapezius (MT), and lower trapezius (LT) muscles during the BSR-SER exercise. Twenty healthy participants will perform the exercise in various lower extremity positions (standing, squat, lunge) and on both stable and unstable surfaces using a BOSU® ball. EMG data will be collected using a wireless surface EMG system and analyzed in terms of percentage of maximal voluntary isometric contraction (%MVIC).

The results of this study may provide valuable insights into the optimization of scapular stabilization exercises and guide clinicians in designing more effective shoulder rehabilitation programs by incorporating kinetic chain principles and unstable surfaces.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years
* Body Mass Index (BMI) less than 30 kg/m²

Exclusion Criteria:

* Engaging in more than 6 hours per week of overhead sports or upper extremity strength training
* History of surgery in the spine, lower extremities, or upper extremities
* Experiencing pain in these regions within the past 6 weeks
* Having a rheumatologic, systemic, or metabolic disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Upper Trapezius Muscle Activation | Day 1 (during the exercise session)
  Surface electromyography (EMG) will measure the muscle activation level of the upper trapezius during the stationary phase of the BSR-SER exercise under various conditions. The activation will be normalized as a percentage of maximal voluntary isometric contraction (%MVIC).
Middle Trapezius Muscle Activation | Day 1 (during the exercise session)
  Surface EMG will measure the muscle activation level of the middle trapezius muscle during the stationary phase of the BSR-SER exercise under different surface and lower limb position conditions. Activation levels will be expressed as %MVIC.
Lower Trapezius Muscle Activation | Day 1 (during the exercise session)
  Surface EMG will measure the muscle activation of the lower trapezius during the stationary phase of the BSR-SER exercise. Muscle activity will be normalized to %MVIC.
Muscle Activation Ratios | Day 1 (during the exercise session)
  Ratios of muscle activation between the upper, middle, and lower trapezius muscles will be calculated to assess balance of muscle recruitment during exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Cobanoglu Demirkan, PhD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colado JC, Garcia-Masso X, Triplett NT, Calatayud J, Flandez J, Behm D, Rogers ME. Construct and concurrent validation of a new resistance intensity scale for exercise with thera-band(R) elastic bands. J Sports Sci Med. 2014 Dec 1;13(4):758-66. eCollection 2014 Dec. PMID 25435767
- [Background] Ecemis ZB, Cobanoglu G, Oksuz BS, Kaya B, Guzel NA, Kafa B, Kafa N. Trapezius Muscle Electromyographic Activity in Lawn-Mower Exercise: Standing Versus Quadruped. J Sport Rehabil. 2024 Dec 10;34(4):436-442. doi: 10.1123/jsr.2023-0404. Print 2025 May 1. PMID 39657698
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Background] Cobanoglu G, Guzel NA, Ecemis ZB, Demirkan MY. Investigation of muscle activation during kinetic chain based exercises in individuals with and without forward head posture. J Back Musculoskelet Rehabil. 2024;37(6):1537-1549. doi: 10.3233/BMR-230397. PMID 38968043
- [Background] Kara D, Harput G, Duzgun I. Trapezius muscle activation levels and ratios during scapular retraction exercises: A comparative study between patients with subacromial impingement syndrome and healthy controls. Clin Biomech (Bristol). 2019 Jul;67:119-126. doi: 10.1016/j.clinbiomech.2019.05.020. Epub 2019 May 11. PMID 31103961
- [Background] Melo ASC, Vilas-Boas JP, Cruz EB, Macedo RM, E Ferreira SB, Sousa AS. The influence of shoulder position during multi-joint exercises in the relative scapular muscles activity in symptomatic and asymptomatic conditions. J Back Musculoskelet Rehabil. 2023;36(4):883-893. doi: 10.3233/BMR-220056. PMID 36776036
- [Background] Uysal O, Akoglu AS, Kara D, Sezik AC, Calik M, Duzgun I. Theraband Applications for Improved Upper Extremity Wall-Slide Exercises. J Athl Train. 2022 Aug 1;57(8):795-803. doi: 10.4085/1062-6050-0305.21. PMID 36356616
- [Background] Mendez-Rebolledo G, Morales-Verdugo J, Orozco-Chavez I, Habechian FAP, Padilla EL, de la Rosa FJB. Optimal activation ratio of the scapular muscles in closed kinetic chain shoulder exercises: A systematic review. J Back Musculoskelet Rehabil. 2021;34(1):3-16. doi: 10.3233/BMR-191771. PMID 32831190